CLINICAL TRIAL: NCT06167369
Title: Biological and Cognitive Marker of Neurodegeneration in Obstructive Sleep Apnea Patients
Status: Recruiting | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Responsible Party: Principal Investigator, Tony Sehr, Principal Investigator, Technische Universität Dresden
Other Study IDs: MeDDrive: BICONOS
Record Dates: First submitted 2023-11-23; First posted 2023-12-12 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Sleep Apnea, Obstructive
Keywords: Sleep apnea; Neurodegeneration; Neurofilament light chain; Glial fibrillary acidic protein; Positive airway pressure therapy
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes; Nerve Degeneration; Charcot-Marie-Tooth disease, Type 1F

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum samples for measurement of neurobiological parameters like Neurofilament light chain or Glial fibrillary acidic protein
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Newly diagnosed sleep apnea patients, starting clinical prescribed positive airway pressure therapy

SUMMARY:
The goal of this observational study is to investigate biomarkers and neurocognitive markers of neurodegenerative processes in obstructive sleep apnea patients.

The main questions the study aims to answer are:

* Does neurodegeneration assessed by neurobiological markers and neurocognitive test performance exists in obstructive sleep apnea?
* Are these neurodegenerative markers are associated with the adherence to clinical prescribed positive airway pressure therapy?

Newly diagnosed patients with obstructive sleep apnea will be observed during the use of clinical prescribed positive pressure therapy. Different study related investigations take place before and six months after treatment start.

Researchers will compare after six months the group of adherent treatment participants with the non-adherent treatment participants group to investigate if differences in the observed neurobiological or neurocognitive parameters exist.

ELIGIBILITY:
Inclusion Criteria:

* newly diagnosed obstructive sleep apnea
* clinical indication for start of positive airwas pressure therapy
* Age older than 18 years

Exclusion Criteria:

* neurodegenerative disease
* Multiple sclerosis
* Stroke within last 3 months
* Brain injury within last 3 months
* MoCA < 21 points
* higher degree chonic kidney disease (lower than 30 mL/min)
* regular use of sleep pills (e.g. Zopiclon, Mirtazapin, Daridorexant)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that are reffered to the sleep lab of the University Hospital Dresden
Sampling Method: Non-Probability Sample
Enrollment: 136 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Concentration of neurofilament light chain | From enrollment to the follow up time point after 6 months of treatment
  longitudinal analysis

SECONDARY OUTCOMES:
Concentration of Neurofilament light chain | From enrollment to the follow up time point after 6 months of treatment, in between the groups
  in between the groups (assessed after 6 months)
Concentration of Glial fibrillary acidic protein | From enrollment to the follow up time point after 6 months of treatment
  longitudinal analysis and in between the groups (assessed after 6 months)
Cognitive performance measured by SDMT, MoCA | From enrollment to the follow up time point after 6 months of treatment
  Longitudinal analysis and in between the groups (assessed after 6 months)
Objective sleep parameters measured by polysomnography or equivalent measuremt methods | From enrollment to the follow up time point after 6 months of treatment
  Longitudinal analysis and in between the groups (assessed after 6 months). For example objective parameters like apnea-hypopnea-index per hour or sleep efficacy in %.
Subjective sleep parameters measured by symptoms questionnaires (Epworth Sleepiness Scale, Pittsburgh Sleep Quality Index) | From enrollment to the follow up time point after 6 months of treatment
  Longitudinal analysis and in between the groups (assessed after 6 months). For example parameters like sleepiness (ESS-questionnnaire, min to max 0 to 24 points) or sleep quality (PSQI-questionnaire, min to max 0 to 21 points). Lower score values represent fewer symptom load.

CONTACTS AND LOCATIONS:
Locations (1):
- Technische Universität Dresden, Universitätsklinikum Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No